CLINICAL TRIAL: NCT03348332
Title: Effect of Supervised Exercise During Pregnancy on Maternal and Newborn Intrapartum Health
Brief Title: Effect During Pregnancy and Intrapartum Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, María Perales Santaella, PhD, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Intrapartum assessment
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Pregnancy
Keywords: exercise; intrapartum; aerobic exercise; resistance exercise; wellbeing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary pregnant women (No Intervention): Pregnant women who do not exercise regularly during pregnancy
- Exercise pregnant women (Experimental): Pregnant women who participate in a supervised exercise program
  Interventions: Behavioral: Exercise pregnant women

INTERVENTIONS:
Behavioral: Exercise pregnant women — A supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (from week 10 to 39) was conducted. Each session consisted of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training. Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60 of maximal heart rate. All subjects wore a heart rate (HR) monitor during the training sessions to control the intensity.
  Arms: Exercise pregnant women

SUMMARY:
Assessing the role of moderate exercise in newborn intrapartum variables have showed to be crucial not only on prescribing exercise safely, but also on understanding its impact on the prevention of some cardio-metabolic diseases after labor. Clarify this concept will be essential on reducing human risk for some chronic diseases through implementing supervised exercise programs during such a critical period.

DETAILED DESCRIPTION:
The aim of this randomized controlled trial was to evaluate the effect of combined exercise (aerobic and strength exercise) on maternal and newborn intrapartum variables.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines.
* Being able to communicate in spanish
* Giving birth at Hospital Universitario de Puerta de Hierro (Majadahonda); Hospital Universitario Severo Ochoa (Leganés).

Exclusion Criteria:

* Multiparity
* Obstetrician complications
* Being interested in the study after 18 weeks
* Not being regular in physical exercise program
* Younger than 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 530 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Stage of labor | At the moment of delivery
  Duration stages of labor (min)

SECONDARY OUTCOMES:
Maternal gestational weight gain | 40-42 weeks of gestation
  Change from baseline in maternal gestational weight gain (g)
Glucose state | 24-26 weeks of gestation
  Maternal glucose state (O´Sullivan test)
Blood pressure | 12, 20 and 34 weeks of gestation
  Maternal blood pressure during pregnancy (mmHg)
Gestational age | At the moment of delivery
  Gestational age (weeks)
Birth weight | At the moment of delivery
  Newborn weight (g)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat Carballo, PhD, Study Director — Universidad Politecnica de Madrid; María Perales Santaella, PhD, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Spain